CLINICAL TRIAL: NCT05552872
Title: A Multicenter Clinical Study on Diagnosis Value of mNGS Technology Among Diabetic Patients With Pulmonary Infections
Brief Title: Study on Diagnosis Value of mNGS Technology Among Diabetic Patients With Pulmonary Infections
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, ZHOU Min, Chief Physician of Department of Respiratory Medicine, Ruijin Hospital
Other Study IDs: 2022Ultra
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus; Pulmonary Infection
Keywords: Pulmonary Infection; Diabetes Mellitus; mNGS; host immune response
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulmonary Infection with DM group: Patients with diabetes and pulmonary infection
  Interventions: Diagnostic Test: mNGS, IDSeq UltraTM
- Pulmonary Infection group: Patients with pulmonary infection while the fasting blood-glucose in the normal range.
  Interventions: Diagnostic Test: mNGS, IDSeq UltraTM

INTERVENTIONS:
Diagnostic Test: mNGS, IDSeq UltraTM — pathogen detection

SUMMARY:
Focusing on patients with diabetes complicated with pulmonary infection, the purpose of this study is: 1) to identify the epidemiology, etiologic spectrum and status of diagnosis and treatment; 2) to explore the lower respiratory microenvironment and host immune response and then make an application in clinic.

DETAILED DESCRIPTION:
Investigators perform a cross-sectional multicenter study on patients with pulmonary infection. All patients receive clinical questionnaires, laboratory examinations and treatment monitoring. Routine clinical pathogen culture and mNGS are both carried out on pathogen detection. Among participants in IDSeq UltraTM group, 1:2 nested case-control study is carried out involving 77 cases from pulmonary-infected group paired with 154 control cases and peripheral blood RNA-seq is carried out between pneumonia patients with diabetes and pneumonia patients without diabetes matched for gender, age and fasting blood-glucose.

The final purpose is to find out the difference in etiologic spectrum and host immune on lower respiratory infection between diabetes patients and controls. Now investigators wish to register this study to do a further research, in order to improve the diagnosis value of diabetes complicated with pulmonary infection and to reduce the mortality.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis by pathogen examination: positive
* Diagnosis through X-ray or CT: characteristic features of pulmonary infection
* Age older than 18 years

Exclusion Criteria:

* Irregular follow-up and lost follow-up
* Withdraw from the study for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Diagnosis by pathogen examination: positive
  * Diagnosis through X-ray or CT: characteristic features of pulmonary infection
  * Age older than 18 years
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Survival at 28 Days | 28 days from date of diagnosis of pulmonary infection until the date of death from any cause, whichever came first
  28 days from date of diagnosis of pulmonary infection until the date of death from any cause
Survival at 14 Days | 14 days from date of diagnosis of pulmonary infection until the date of death from any cause, whichever came first
  14 days from date of diagnosis of pulmonary infection until the date of death from any cause
Survival at 7 Days | 7 days from date of diagnosis of pulmonary infection until the date of death from any cause, whichever came first
  7 days from date of diagnosis of pulmonary infection until the date of death from any cause

SECONDARY OUTCOMES:
72h Treatment Response | disease treating 72 hours
  response after infection treating 72 hours
Hospitalization Time | Every 6 months from date of diagnosis of pulmonary infection until the date of death from any cause, assessed up to 3 years
  the time of hospital stay including ordinary sickroom and ICU of patients from different groups
CURB-65 Score | Every 6 months from date of diagnosis of pulmonary infection until the date of death from any cause, assessed up to 3 years
  Differences in confusion, urea, respiratory rate and age 65 scoring system from different groups.
Inflammatory Parameters | Day 0, day 3, day7-14 and final result from date of diagnosis of pulmonary infection until the date of death or cure from any cause, assessed up to 1 years
  Differences in CRP, PCT, IL-6, IL-8, TNF-α from different groups.
Cell-mediated Immunoserologic Indexs | Day 0, day 3, day7-14 and final result from date of diagnosis of pulmonary infection until the date of death or cure from any cause, assessed up to 1 years
  Differences of CD3, CD4 and CD8 in different groups in order to research on cell-mediated immunity of patients with or without diabetes and pulmonary infection
PSI Indexs | Day 0, day 3, day7-14 and final result from date of diagnosis of pulmonary infection until the date of death or cure from any cause, assessed up to 1 years
  Pneumonia severity index grade, including age, comorbidities, signs, blood gases
SOFA Indexs | Day 0, day 3, day7-14 and final result from date of diagnosis of pulmonary infection until the date of death or cure from any cause, assessed up to 1 years
  Sequential Organ Failure Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jieming Qu, Ph.D., M.D., Principal Investigator — China, Shanghai Ruijin Hospital Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No